CLINICAL TRIAL: NCT06300814
Title: The Effect of Progressive Relaxation Exercise and Music Recital on Sleep, Quality of Life and Emotional State in Children With Epilepsy
Brief Title: The Effect of Exercise and Music on Sleep, Quality of Life and Emotional State in Children With Epilepsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Emre Usta, Research Assistant, TC Erciyes University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: ERU-HEM-EU-01
Record Dates: First submitted 2024-03-01; First posted 2024-03-08 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Epilepsy in Children
Keywords: Exercise; Music; Sleep; Quality of life
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Progressive relaxation exercise group (Experimental): 15 children aged 9-16 years who met the inclusion and exclusion criteria.
  Interventions: Other: Progressive relaxation exercise group
- Music recital group (Experimental): 15 children aged 9-16 years who met the inclusion and exclusion criteria.
  Interventions: Other: Music recital group
- Control group (No Intervention): 15 children aged 9-16 years who met the inclusion and exclusion criteria.

INTERVENTIONS:
Other: Progressive relaxation exercise group — A video containing the progressive relaxation exercise was sent to the phones of the mothers of children diagnosed with epilepsy in the intervention group to whom progressive relaxation exercise would be applied, and the children applied progressive relaxation exercise (15 minutes of progressive relaxation exercise before bedtime for a total of 4 weeks, 5 days a week).
  Arms: Progressive relaxation exercise group
Other: Music recital group — The link of the music recital (link) was sent to the phones of the mothers of children diagnosed with epilepsy in the intervention group, where the music concert will be applied, and the children listened to it (music concert was applied for 15 minutes before going to bed, 5 days a week for a total of 4 weeks).
  Arms: Music recital group

SUMMARY:
This study was planned as a randomized controlled experimental study with a pretest-posttest design to determine the effect of parental supervision and video-guided progressive relaxation exercise (PRE) and music recital on sleep, quality of life and emotional states in children with epilepsy aged 9-16 years. The main questions it aims to answer are as follows:

According to the evaluation of children with epilepsy, does the progressive relaxation exercise applied to children have an effect on sleep, quality of life and emotional states? According to the evaluation of children with epilepsy, does music recital applied to children have an effect on sleep quality of life and emotional states? The study consisted of 45 children (15 children in the progressive relaxation exercise group, 15 children in the music recital group and 15 children in the control group). Ethics committee approval, permission from the institutions and informed consent of the children were obtained for the conduct of the study. A value of p<0.05 was considered statistically significant in data analysis.

DETAILED DESCRIPTION:
This randomized controlled experimental study will be conducted to evaluate the effect of progressive relaxation exercise and music recital before going to sleep on sleep, quality of life and emotional state in children with epilepsy. The study will be conducted with children aged 9-16 years and their mothers hospitalized in a tertiary care hospital. Children in the progressive relaxation exercise (n=15), music recital (n=15) and control (n=15) groups will be selected similarly in terms of age, gender, educational status, duration of diagnosis and number. The data of the study will be collected with the Quality of Life Scale in Children Parent Form (QoLQS-PPP), Pediatric Symptom Checklist-17 (PSCL-17), Child Sleep Habits Questionnaire (CSHQ) to be administered to mothers and the Quality of Life Scale in Children Child and Adolescent Form (QoLQ-C), Me and My Emotions in Children and Adolescents Scale (MEAS), and Sleep Deprivation Scale for Children and Adolescents (PSSAD) to be administered to children. Children in the PRE group will be asked to do PRE before going to sleep five days a week (4 weeks) with a PRE video for a total of 15 minutes each session. Children in the music group will be asked to listen to the selected music before going to sleep five days a week (4 weeks) for a total of 15 minutes each session. These scales will be applied to the children before the interventions (Time 1). After the interventions were performed five days a week (4 weeks) for a total of 15 minutes each session before going to sleep, the same scales will be applied again (Time 2) and the results of the study will be compared. Children in the control group will receive standard treatment. In the evaluation of the data showing normal distribution; Student t (between 2 groups) and One Way ANOVA (more than 2 groups) tests will be used to test whether there is a difference between two independent groups; Paired-samples t test will be used to test whether there is a difference between the measurements before and after the intervention. In the evaluation of non-normally distributed data; Mann-Whitney U (between 2 groups) and Kruskal-Wallis Analysis of Variance (more than 2 groups) tests will be used to test whether there is a difference between two independent groups; Wilcoxon Paired-Samples Test will be used to test whether there is a difference between pre and post intervention measurements. A value of p<0.05 was considered statistically significant in data analysis.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 9-16,
* Does not have a chronic or genetic disease other than epilepsy,
* No mental, visual or hearing impairment,
* Having a mother who is at least a primary school graduate,
* Both he and his mother are open to communication and cooperation,
* Children who both themselves and their mothers volunteer to participate in the research and give verbal and written consent.

Exclusion Criteria:

* Not between the ages of 9-16,
* Having a chronic or genetic disease other than epilepsy,
* Mentally, visually or hearing impaired,
* Mothers who are not primary school graduates,
* Both he and his mother are not open to communication and cooperation,
* Neither they nor their mothers volunteered to participate in the research,
* Children and mothers without smart phones

Ages: 9 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 45 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2025-03-26 (Actual)

PRIMARY OUTCOMES:
The Children's Sleep Habits Questionnaire (CSHQ) | Average 30 days: pre-intervention measurement (Time 1), 4 weeks intervention, immediately after the intervention measurement (Time 2)
  CSHQ, which consists of 8 subscales (resistance to going to bed, difficulty sleeping, total sleep time, sleep anxiety, frequent waking up at night, sleepiness during the day, breathing-related sleep problems and parasomnia) and 33 items, is scored 1-3 points (1 = rarely…. 3 = It is generally evaluated as).

SECONDARY OUTCOMES:
The Pediatric Quality of Life Inventory (PedsQL) | Average 30 days: pre-intervention measurement (Time 1), 4 weeks intervention, immediately after the intervention measurement (Time 2)
  Scale; It consists of 23 items in total: physical health = 8, emotional functionality = 5, social functionality = 5, school functionality = 5 items. The same items are available in all child and parent forms created according to age groups. When answering the scale, a score of 0-4 was determined for each question (0 = never… 4 = almost always).
The Me and My School Questionnaire (M&MS) | Average 30 days: pre-intervention measurement (Time 1), 4 weeks intervention, immediately after the intervention measurement (Time 2)
  It consists of a total of 16 items: emotional difficulties = 10, behavioral problems = 6 items. Each item in the scale; It evaluates to never = 0, sometimes = 1, always = 2. High scores on each subscale indicate the likelihood of mental health problems

CONTACTS AND LOCATIONS:
Overall Officials: Emre Usta, Principal Investigator — TC Erciyes University
Locations (1):
- Erciyes University, Kayseri, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No